CLINICAL TRIAL: NCT01152983
Title: Single Center, Open Label, Prospective, Non-comparative, Non-randomized Study to Assess the Safety and Performance of the Rapid Ring Device (Comparative Study to Assess the Pain Reduction)
Brief Title: Safety and Performance Evaluation of the Rapid Ring Device
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RapiDx Ltd. (Industry)
Responsible Party: Erez Rozenfeld, RapiDx Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTIL - CL-001
Record Dates: First submitted 2010-06-27; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Finger sticks; Rapid Ring; Finger sticks method of obtaining blood for diagnostic testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Rapid Ring — Rapid Ring is a ring-shaped device that encircles the distal phalanx of the middle finger and blocks the arterial blood to quickly and passively withdraw blood following a finger stick, and to reduce the pain of the lancet.

SUMMARY:
The purpose of this study is to demonstrate the safety, performance and initial efficacy of the RapiDx device.

DETAILED DESCRIPTION:
The study will be a single center, open label, prospective, non-comparative, randomized trial and assess the safety and performance of the Rapid Ring device. In order to assess pain reduction, a comparative study will be performed and each subject will serve as his/her own control.

Clinical assessment for all 100% patients will occur at baseline. All participants will be men and women above the age of 18. The trial will be conducted at a Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy
* Subject's age is between 18 to 70 years old
* Subject must be capable of providing informed consent

Exclusion Criteria:

* Clotting disorders
* Subject has a clinically significant untreated chronic disease which may unable him/ her to participate in the study.
* Subject is taking anti-coagulant medication
* Non-intact finger tip (left middle/ring finger)
* Skin disease on the subject finger
* Abnormal blood pressure
* Pregnant or lactating women
* Menstrual period
* Previous diagnosis of HIV or Hepatitis
* Participation in other clinical investigations within previous 30 days
* Peripheral blood vessels diseases
* Diabetes
* Neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Collection of at least 2 drops (approximately 50microliter) of blood within one minute. | approximately 6 months

SECONDARY OUTCOMES:
Reduction in pain | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ella Naparstek, Prof., Principal Investigator — Chairman of the Hematology Institute and the Department of Hematology and Bone Marrow Transplantation at Tel Aviv Sourasky Medical Center.
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel